CLINICAL TRIAL: NCT02918786
Title: The Efficacy of the Whisperflow CPAP System Versus High Flow Nasal Cannula Oxygen Therapy in Patients at High Risk for Postextubation Failure
Brief Title: The Efficacy of the Whisperflow CPAP System Versus Nasal High Flow in Patients at High Risk for Postextubation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Pongdhep Theerawit, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID 12-58-11
Record Dates: First submitted 2016-08-16; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Respiratory Failure
Keywords: oxygen therapy; continuous positive airway pressure; extubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous positive airway pressure (Active Comparator): After extubation, patients will receive continuous positive airway pressure (CPAP) delivered by the variable generator WhisperFlow System (control) Intervention:Device : CPAP of 5 cmH2O delivered by the variable generator WhisperFlow System for 48 hours
  Interventions: Device: CPAP
- Nasal high-flow (Active Comparator): After extubation, patients will receive oxygen therapy through the nasal high-flow (intervention) Intervention: Device: Nasal high-flow
  Interventions: Device: Nasal high-flow

INTERVENTIONS:
Device: Nasal high-flow — After extubation, the patients will receive oxygen delivered through the nasal high-flow system (Optiflow™). The FiO2 will be adjusted in order to obtain a SpO2 between 92% and 98% in hypoxemic patients and between 88% and 95% in hypercapnic patients. Gas flow will be set until maximal level of 60 LPM.
  Arms: Nasal high-flow
Device: CPAP — After extubation, patients will receive CPAP at 5 cmH2O delivered by the variable generator WhisperFlow System. The FiO2 will be adjusted in order to obtain a SpO2 between 92% and 98% in hypoxemic patients and between 88% and 95% in hypercapnic patients.
  Arms: Continuous positive airway pressure

SUMMARY:
The purpose of this study is to compare the effect of continuous positive airway pressure (CPAP) delivered by the variable generator WhisperFlow System with high flow nasal cannula oxygen therapy in mechanically ventilated patient who are at risk for postextubation failure.

DETAILED DESCRIPTION:
Postextubation respiratory failure is not an uncommon condition after discontinuation of mechanical ventilation. Subsequently reintubation and mechanical ventilation for postextubation respiratory failure may lead to increasing of hospital morbidity and mortality and and prolonging intensive care and hospital stay. Several studies have demonstrated the efficacy of non-invasive ventilation to prevent the postextubation failure in patients with high risk for extubation failure.

The variable generator whisper flow system ((Philips Respironics, Murrysville, PA, USA) is the one of widely used continuous positive airway pressure(CPAP) device in UK. This device employs an oxygen-driven venturi to entrain air and generates high fresh gas flow up to 140 liter per minute. The oxygen/air mixture enters the breathing circuit and exits through a threshold resistor namely CPAP valve. Whisperflow is able to provide the flow into the breathing system via oronasal mask which exceeds the peak inspiratory flow rate of the patient and may improve work of breathing as well as gas exchange. In daily clinical practice, the investigators apply this device with humidifier in patients with weaning difficulty and patients who are at risk for postextubation failure.

High-flow nasal oxygen therapy(HFNO) is a device which heated and humidified oxygen is distributed to the nose at high flow rates. With the high flow rate (up to 60 Liter per minute), it generates low level of positive airway pressure. Physiological benefits of HFNO comprises decreasing of the dead space, work of breathing and the low level of positive airway pressure associated with better lung recruitment. Furthermore, the fraction of inspired oxygen can be adjusted and measured by changing the fraction of oxygen in the driving gas.

In the present randomized, controlled trial, the investigators will compare two devices for oxygen therapy, with low levels of continuous positive airway pressure, nasal high-flow oxygen therapy and CPAP of 5 cmH2O delivered by the variable generator WhisperFlow System with oronasal mask , in critically ill patients who are at risk for postextubation failure. The investigators hypothesize that nasal high-flow is superior to CPAP the in terms of reintubation rate.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation > 48 hours and
* high risk for extubation failure namely , congestive heart failure, ineffective cough and excessive tracheobronchial secretions, more than one failure of a weaning trial, more than one co-morbid condition, patients who had hypercapnia, and upper airway obstruction without immediately required intubation

Exclusion Criteria:

* age<18 years
* pregnancy
* tracheostomy
* uncontrolled cardiac ischemia or arrhythmias
* unstable hemodynamic status
* documented swallowing problem
* documented cervical spine injury
* Facial anatomical abnormalities interfering with the mask fit
* agitated or uncooperative state
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Reintubation rate | 48 hours
  Number of participants who required reintubation within 48 hours after extubation

SECONDARY OUTCOMES:
post extubation respiratory failure | 48 hours
  Number of participants who required either reintubation or application of Bi-level noninvasive positive airway pressure within 48 hours after extubation

OTHER OUTCOMES:
Length of ICU stay | 30 days
Patient's discomfort | 48 hours
  The investigators will assessed the discomfort of participants by Critical-Care Pain Observation Tool.
oxygen desaturations | 48 hours
  The participants will be monitored and recorded oxygen saturation with the pulse oximeter at 15 minutes, 2 hours, 24 hours and 48 hours after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Nava S, Gregoretti C, Fanfulla F, Squadrone E, Grassi M, Carlucci A, Beltrame F, Navalesi P. Noninvasive ventilation to prevent respiratory failure after extubation in high-risk patients. Crit Care Med. 2005 Nov;33(11):2465-70. doi: 10.1097/01.ccm.0000186416.44752.72. PMID 16276167
- [Background] Glover GW, Fletcher SJ. Assessing the performance of the Whisperflow continuous positive airway pressure generator: a bench study. Br J Anaesth. 2009 Jun;102(6):875-81. doi: 10.1093/bja/aep077. Epub 2009 Apr 19. PMID 19380311
- [Background] Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standard weaning criteria. Am J Respir Crit Care Med. 2000 May;161(5):1530-6. doi: 10.1164/ajrccm.161.5.9905102. PMID 10806150
- [Background] Nava S, Hill N. Non-invasive ventilation in acute respiratory failure. Lancet. 2009 Jul 18;374(9685):250-9. doi: 10.1016/S0140-6736(09)60496-7. PMID 19616722